CLINICAL TRIAL: NCT01786096
Title: A Phase 1, Open-Label, Dose-Escalation Study of SGN-CD19A in Patients With B-Lineage Acute Lymphoblastic Leukemia and Highly Aggressive Lymphomas
Brief Title: A Safety Study of SGN-CD19A for Leukemia and Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN19A-001
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Burkitt Lymphoma; Precursor B-cell Lymphoblastic Leukemia-Lymphoma
Keywords: Burkitt Lymphoma; Antibodies, Monoclonal; Antibody-Drug Conjugate; B-Lineage Acute Lymphoblastic Leukemia; B-Lineage Lymphoblastic Lymphoma; Burkitt Leukemia; Monomethylauristatin F; Antigens, CD19; Drug Therapy
MeSH Terms: conditions — Burkitt Lymphoma; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SGN-CD19A (Experimental): SGN-CD19A (IV) once (Day 1) or twice (Days 1 and 8) every 21 days; dose range: 0.3-6 mg/kg
  Interventions: Drug: SGN-CD19A

INTERVENTIONS:
Drug: SGN-CD19A — SGN-CD19A (IV) once (Day 1) or twice (Days 1 and 8) every 21 days; dose range: 0.3-6 mg/kg

SUMMARY:
This is a phase 1, open-label, dose-escalation, multicenter study to evaluate the safety and tolerability of SGN-CD19A in adult and pediatric patients with relapsed or refractory B-lineage acute lymphoblastic leukemia (B-ALL), Burkitt lymphoma or leukemia, or B-lineage lymphoblastic lymphoma (B-LBL).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients must be relapsed or refractory to at least 1 prior multi-agent systemic therapy. Pediatric patients must be relapsed or refractory to at least 2 prior multi-agent systemic therapies. Patients with acute lymphoblastic leukemia who are Philadelphia chromosome-positive must have failed a second generation tyrosine kinase inhibitor.
* Eastern Cooperative Oncology Group status of 2 or lower
* Pathologically confirmed diagnosis of B-lineage acute lymphoblastic leukemia, Burkitt leukemia or lymphoma, or B-lineage lymphoblastic lymphoma
* Measurable disease

Exclusion Criteria:

* Allogeneic stem cell transplant within 60 days, active acute or chronic graft-versus-host disease (GvHD), or receiving immunosuppressive therapy as treatment for GvHD

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-02; Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Through 1 month post last dose
Incidence of laboratory abnormalities | Through 1 month post last dose

SECONDARY OUTCOMES:
Objective response according to modified response criteria for acute myeloid leukemia (Cheson 2003) or revised response criteria for malignant lymphoma (Cheson 2007) | Through 1 month post last dose
Duration of response | Until disease progression or start of new anticancer treatment, an expected average of 3 months
Overall survival | Until death or study closure, an expected average of 6 months
Blood concentrations of SGN-CD19A and metabolites | Cycles 1, 2, and 4: predose, 30 minutes, and up to 2, 4, 8, 24, 72, 120, 168, and 336 hours post dose start; All other cycles: predose, 30 minutes, and 168 and 336 hours post dose start; and 1 month post last dose
Incidence of antitherapeutic antibodies | Predose in most cycles and 1 month post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Eric Feldman, MD, Study Director — Seagen Inc.
Locations (13):
- United States (13):
  - Children's Hospital of Alabama / University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Children's Healthcare of Atlanta / Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio